CLINICAL TRIAL: NCT04236908
Title: Accessible Acupuncture for the Warrior With Acute Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: David Moss (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, David Moss, Principal Investigator, Mike O'Callaghan Military Hospital
Organization: Mike O'Callaghan Military Hospital (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FWH20200025H
Record Dates: First submitted 2020-01-17; First posted 2020-01-22 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Acupuncture; Low Back Pain
Keywords: acupuncture; low back pain
MeSH Terms: conditions — Low Back Pain | interventions — Anti-Inflammatory Agents, Non-Steroidal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (4):
- Group 1 (NSAIDS only) (Experimental): NSAIDs only (naproxen 500mg by mouth twice a day as needed)
  Interventions: Drug: NSAIDS
- Group 2 (Acupuncture+GV26) (Experimental): Acupuncture to include use of GV 26 with manual tonification (twisting or rotating the needle) plus NSAIDs (naproxen 500mg by mouth twice a day as needed)
  Interventions: Drug: NSAIDS; Device: GV26 with manual tonification
- Group 3 (Battlefield Acupuncture+NSAIDS) (Experimental): Battlefield Acupuncture in both ears (which includes the points cingulate gyrus, thalamus, omega-2, point zero and shen men) plus NSAIDs (naproxen 500mg by mouth twice a day as needed)
  Interventions: Drug: NSAIDS; Device: Battlefield Acupuncture
- Group 4 (Battlefield Acupuncture+GV26+NSAIDS) (Experimental): GV26 with manual tonification + Battlefield Acupuncture in both ears (which includes the points cingulate gyrus, thalamus, omega-2, point zero and shen men) plus NSAIDs (naproxen 500mg by mouth twice a day as needed).
  Interventions: Drug: NSAIDS; Device: Battlefield Acupuncture; Device: GV26 with manual tonification

INTERVENTIONS:
Drug: NSAIDS — Naproxen 500mg by mouth twice a day as needed.
Device: Battlefield Acupuncture — Battlefield Acupuncture in both ears (which includes the points cingulate gyrus, thalamus, omega-2, point zero and shen men).
  Battlefield acupuncture utilizes up to 10 ASP acupuncture needles (5 in each ear). The Battlefield Acupuncture points include: cingulate gyrus, thalamus, omega-2, point zero, and shen men. The semi-permanent needles are left in place and typically stay in place for 2-7 days. Needles will usually fall out on their own, can be removed by the patient or the patient can call study staff and come in for removal if desired.
  Arms: Group 3 (Battlefield Acupuncture+NSAIDS); Group 4 (Battlefield Acupuncture+GV26+NSAIDS)
Device: GV26 with manual tonification — Acupuncture to include use of GV 26 with manual tonification (twisting or rotating the needle).
  The protocol for using GV26 is as follows: With the patient in a seated position the acupuncturist places a 40mm needle in the acupuncture point GV26 (located on the philtrum, on the anterior midline, at the junction of the upper 1/3 and lower 2/3 of the distance from the nose to the margin of the upper lip). The acupuncturist then rapidly rotates the needle at the handle clockwise and counterclockwise (known as manual tonification) for 20-40 seconds at a time. The patient then stands up and assesses their pain. This will be performed up to 6 cycles. If a patient is unable to sit or stand, this may also be performed in a supine position with the patient attempting to sit or stand every 20-40 seconds.
  Arms: Group 2 (Acupuncture+GV26); Group 4 (Battlefield Acupuncture+GV26+NSAIDS)

SUMMARY:
The objective of this study is to determine if auricular acupuncture and/or the acupuncture point governor vessel 26 (GV26) with manual tonification is superior to conservative management (NSAIDs) at reducing acute low back pain (less than 4 weeks in duration).

DETAILED DESCRIPTION:
The study will be a randomized control trial of Active Duty and DoD Beneficiaries aged 18 years or older with complaints of acute lower back pain (four weeks or less in duration). Subjects will be randomized into one of four study groups receiving either 1) NSAIDs only (naproxen 500mg by mouth twice a day as needed) or 2) acupuncture to include use of GV 26 with manual tonification (twisting or rotating the needle) plus NSAIDs (naproxen 500mg by mouth twice a day as needed) or 3) Battlefield Acupuncture in both ears (which includes the points cingulate gyrus, thalamus, omega-2, point zero and shen men) plus NSAIDs (naproxen 500mg by mouth twice a day as needed) or 4) GV26 with manual tonification + Battlefield Acupuncture in both ears (which includes the points cingulate gyrus, thalamus, omega-2, point zero and shen men) plus NSAIDs (naproxen 500mg by mouth twice a day as needed). We seek to determine if acupuncture is superior to conservative management alone in treating acute low back pain (4 weeks or less in duration).

ELIGIBILITY:
**Patients must be able to get care at Nellis Air Force Base (a military installation) in order to participate in this study**

Inclusion Criteria:

* Male and Female Active Duty and DoD Beneficiaries aged 18 years or older.
* Complaints of acute back pain (4 weeks or less in duration).

Exclusion Criteria:

* Known history of underlying rheumatologic condition.
* Chronic low back pain (greater than 4 weeks in duration).
* Contraindications to NSAID use (including peptic ulcer disease, underlying coagulopathy, severe coronary artery disease, underlying renal disease, allergy, thrombocytopenia).
* Red flag symptoms of low back pain (to include bowel or bladder incontinence, sudden onset sensorineural deficits, loss of sensation in the perineal region).
* Requiring narcotic use to control symptoms.
* Patients currently taking opioid medications.
* pregnant, may be pregnant, or attempting to become pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 276 (Actual)
Dates: Start 2020-08-25 (Actual); Primary Completion 2025-12-09 (Actual); Study Completion 2025-12-09 (Actual)

PRIMARY OUTCOMES:
Change in Defense and Veterans Pain Rating Scale (DVPRS) | Pre-treatment: time 0 (week 1); post-treatment (week 2 followup)
  The DVPRS consists of an 11-point numerical rating scale with 0 indicating no pain and 10 indicating severe pain. It has been confirmed for reliability and validity in measuring both acute and chronic pain, and is currently the standard for pain measurement throughout DoD and VA health systems. The DVPRS has demonstrated linear scale qualities allowing parametric methods to be used.
Number of days missed from work due to lower back pain. | Post-treatment (Visit 2, 1 week followup)
  The number of days missed from work is self-explanatory and will be treated as a parametric interval variable.

CONTACTS AND LOCATIONS:
Locations (1):
- Mike O'Callaghan Military Medical Center, Nellis Air Force Base, Nevada, United States

IPD SHARING:
Plan to Share IPD: No
We do not plan on sharing data.

REFERENCES:
- [Background] Armed Forces Health Surveillance Branch. Absolute and relative morbidity burdens attributable to various illnesses and injuries, active component, U.S. Armed Forces, 2015. MSMR. 2016 Apr;23(4):2-7. No abstract available. PMID 27152681
- [Background] Armed Forces Health Surveillance Branch. Absolute and relative morbidity burdens attributable to various illnesses and injuries, active component, U.S. Armed Forces, 2016. MSMR. 2017 Apr;24(4):2-8. No abstract available. PMID 28488875
- [Background] Clark LL, Hu Z. Diagnoses of low back pain, active component, U.S. Armed Forces, 2010-2014. MSMR. 2015 Dec;22(12):8-11. PMID 26726722
- [Background] Armed Forces Health Surveillance Center (AFHSC). Medical evacuations from Afghanistan during Operation Enduring Freedom, active and reserve components, U.S. Armed Forces, 7 October 2001-31 December 2012. MSMR. 2013 Jun;20(6):2-8. PMID 23819534
- [Background] Cohen SP, Nguyen C, Kapoor SG, Anderson-Barnes VC, Foster L, Shields C, McLean B, Wichman T, Plunkett A. Back pain during war: an analysis of factors affecting outcome. Arch Intern Med. 2009 Nov 9;169(20):1916-23. doi: 10.1001/archinternmed.2009.380. PMID 19901146
- [Background] Ruscio BA, Jones BH, Bullock SH, Burnham BR, Canham-Chervak M, Rennix CP, Wells TS, Smith JW. A process to identify military injury prevention priorities based on injury type and limited duty days. Am J Prev Med. 2010 Jan;38(1 Suppl):S19-33. doi: 10.1016/j.amepre.2009.10.004. PMID 20117593
- [Background] Liu YT, Chiu CW, Chang CF, Lee TC, Chen CY, Chang SC, Lee CY, Lo LC. Efficacy and Safety of Acupuncture for Acute Low Back Pain in Emergency Department: A Pilot Cohort Study. Evid Based Complement Alternat Med. 2015;2015:179731. doi: 10.1155/2015/179731. Epub 2015 Aug 4. PMID 26346626
- [Background] Knox JB, Orchowski JR, Scher DL, Owens BD, Burks R, Belmont PJ Jr. Occupational driving as a risk factor for low back pain in active-duty military service members. Spine J. 2014 Apr;14(4):592-7. doi: 10.1016/j.spinee.2013.06.029. Epub 2013 Aug 27. PMID 23992937
- [Background] Simon-Arndt CM, Yuan H, Hourani LL. Aircraft type and diagnosed back disorders in U.S. Navy pilots and aircrew. Aviat Space Environ Med. 1997 Nov;68(11):1012-8. PMID 9383501
- [Background] Niebuhr DW, Krampf RL, Mayo JA, Blandford CD, Levin LI, Cowan DN. Risk factors for disability retirement among healthy adults joining the U.S. Army. Mil Med. 2011 Feb;176(2):170-5. doi: 10.7205/milmed-d-10-00114. PMID 21366079
- [Background] Sikorski C, Emerson MA, Cowan DN, Niebuhr DW. Risk factors for medical disability in U.S. enlisted Marines: fiscal years 2001 to 2009. Mil Med. 2012 Feb;177(2):128-34. doi: 10.7205/milmed-d-11-00250. PMID 22360055
- [Background] Holm, S. 1979. A simple sequential rejective multiple test procedure. Scand. J. Statistics, 6: 65-70.
- [Background] R Core Team. R: A language and environment for statistical computing. R Foundation for Statistical Computing, Vienna, Austria. 2016
- [Background] Niemtzow RC. Battlefield Acupuncture: My Story. Med Acupunct. 2018 Apr 1;30(2):57-58. doi: 10.1089/acu.2018.29077.rcn. No abstract available. PMID 29937955